CLINICAL TRIAL: NCT06993688
Title: Revealing Information Genuinely & Honestly Across Time - Communication Preferences Visit (RIGHTimeCPV) Pilot
Brief Title: Revealing Information Genuinely & Honestly Across Time - Communication Preferences Visit
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RIGHTimeCPV; K08CA266935 (NIH); NCI-2025-03410 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2025-05-06; First posted 2025-05-29 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Cancer; Communication
Keywords: Prognostic Communication; Cancer; Poor Prognosis; Participants 12-25 years of age; Caregivers; Pediatric oncologists; Communication Preferences Companions
MeSH Terms: conditions — Neoplasms; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RIGHTimeCPV intervention: Patients and Caregivers (parents) (Other): Pediatric patients aged 12-25 years with poor prognosis cancer who receive treatment at the study site or participating affiliate
  Caregivers of patients of any age who receive treatment at the study site (referred to as 'parent')
  Interventions: Behavioral: Prognostic Communication-Patient/parent
- RIGHTimeCPV intervention: Psychosocial/nursing clinicians (Other): Psychosocial/nursing clinicians who participate in the clinical care of participating patients/parents and serve as communication preferences companions (CPCs) under the auspices of this study
  Interventions: Behavioral: Prognostic Communication-CPC
- RIGHTimeCPV intervention: Pediatric oncologists (Other): Pediatric oncologists who treat participating patients/parents
  Interventions: Behavioral: Prognostic Communication-Oncologist

INTERVENTIONS:
Behavioral: Prognostic Communication-Patient/parent — * Patient/parent identifies and selects a communication preferences companion (CPC)
  * CPC and patient/parent meet for a Communication Preferences Visit (CPV)
  * Oncologist, patient/parent, and CPC attend next disease re-evaluation visit together.
  Arms: RIGHTimeCPV intervention: Patients and Caregivers (parents)
Behavioral: Prognostic Communication-CPC — * CPC reviews intervention materials and conversation guide with the research team
  * CPC and patient/parent meet for a CPV, and CPC documents patient/parent preferences in a templated form
  * CPC and oncologist discuss the CPV form
  * Oncologist, patient/parent, and CPC attend next disease re-evaluation visit together.
  Arms: RIGHTimeCPV intervention: Psychosocial/nursing clinicians
Behavioral: Prognostic Communication-Oncologist — * CPC and oncologist discuss the CPV form
  * Oncologist, patient/parent, and CPC attend next disease re-evaluation visit together
  Arms: RIGHTimeCPV intervention: Pediatric oncologists

SUMMARY:
The purpose of this research study is to obtain insights and feedback from patients and parents about a new approach to support conversations about how cancer may affect one's future life and quality of life (i.e., prognostic communication). This study involves creating a personalized approach to discussing prognosis.

Primary Objectives

* To evaluate the feasibility of implementing the RIGHTimeCPV intervention among pediatric oncology patients, caregivers, and clinicians (referred to herein as "shareholders").
* To assess the acceptability of the intervention across the shareholder groups.

Secondary Objectives

* To explore the potential impact of the RIGHTimeCPV intervention on communication quality, concordance in prognostic understanding, and therapeutic alliance between patients/families and multidisciplinary clinicians.
* To explore whether the practice of eliciting, sharing, and honoring individualized communication preferences is sustained by clinicians after participation in the RIGHTimeCPV intervention.

DETAILED DESCRIPTION:
An estimated range of 52-85 total participants across all subject cohorts at St. Jude and participating affiliate sites, including 12-15 pediatric oncologists, 2-3 family units per participating oncologist (with an emphasis on dyadic recruitment within a given family unit, but also may include independent patients, independent caregivers, or a patient and multiple caregivers; estimated 15-25 patients and 15-25 parents), and 10-20 'communication preferences companions' (CPCs).

The RIGHTimeCPV intervention centers eliciting, sharing, and integrating individualized patient/parent preferences for prognostic communication into routine clinical practice through collaboration between multidisciplinary clinicians on the care team.

The intervention comprises five parts: 1) patient/parent identifies and selects a CPC; 2) CPC reviews intervention materials and conversation guide with the research team; 3) CPC and patient/parent meet for a CPV visit, and CPC documents patient/parent preferences in a templated form; 4) CPC and oncologist discuss the CPV form; 5) oncologist, patient/parent, and CPC attend next disease re-evaluation visit together.

Data will be collected at the following timepoints: 1) study enrollment (routine demographic information collected from each participant); 2) CPV 'conversation guide' training with CPC and research staff (audio-recorded encounter); 3) CPV with patient/parent and CPC (audio-recorded encounter); 4) during the period after a CPV and before the next disease re-evaluation encounter (brief survey and semi-structured interview for patients/parents and oncologists); 5) CPC-oncologist discussion to review the CPV form (email or audio-recorded encounter); 6) disease re-evaluation visit with patient/parent, oncologist, and CPC (audio-recorded encounter); 7) post-intervention interview (brief surveys for patients/parents and oncologists and semi-structured interviews for all participants); and 8) post-intervention interview six months after the final DRV (semi-structured interviews for all participants).

ELIGIBILITY:
Inclusion Criteria: Patients

* Aged 12-25 years diagnosed with poor prognosis cancer (high risk or otherwise difficult to treat cancers), as defined by a pediatric oncologist estimating odds of overall survival as 50% or less
* Anticipated by a pediatric oncologist to have one or more disease re-evaluation timepoints over the next six months
* Not anticipated by a pediatric oncologist to approach end of life in the next three months

Inclusion Criteria: Parents

* Aged 18 years or older and/or legally emancipated
* Parent or other self-identified caregiver of a patient of any age with poor prognosis cancer (as defined above)

Inclusion Criteria: Oncologists

* Pediatric oncologists who treat eligible patients/caregivers at the study site, St. Jude Children's Research Hospital (SJCRH) or its included affiliates:

  * Peoria, IL: The Jim and Trudy Maloof St. Jude Midwest Affiliate Clinic
  * Charlotte, NC: Novant Health Hemby Children's Hospital
  * Shreveport, LA: Ochsner LSU Health-Feist-Weiller Cancer Center

Inclusion Criteria: Communication Preferences Companions (CPCs)

* Multidisciplinary clinicians from a participant's psychosocial or nursing care team, identified by that participant to serve as their 'communication preferences companion' (CPC) during the pilot
* Provides clinical care to pediatric cancer patients under the auspices of psychology, social work, spiritual care, child life, cultural navigation, quality of life/palliative care, or nursing

Exclusion Criteria:

* Does not meet the stated inclusion criteria

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of implementing the RIGHTimeCPV intervention | Between Day 1-30 after a Disease Reevaluation Visit (DRV) [participant specific] and again 6 months after the final DRV during study exit interviews [participant specific
  Quantitative findings of feasibility will be assessed using the Feasibility of Intervention Measure (FIM). The FIM measure includes four itemized responses that are scored from one to five, such that one represents the lowest possible mean score and five the highest possible mean score. Feasibility is standardly considered to be achieved with a mean score ≥3 for this measure. Higher scores indicate greater perceived feasibility of the intervention.
Acceptability of implementing the RIGHTimeCPV intervention | Between Day 1-30 after a Disease Reevaluation Visit (DRV) [participant specific] and again 6 months after the final DRV during study exit interviews [participant specific
  Quantitative findings of acceptability will be assessed using the Acceptability of Intervention Measure (AIM). The AIM measure includes four itemized responses that are scored from one to five, such that one represents the lowest possible mean score and five the highest possible mean score. Acceptability is standardly considered to be achieved with a mean score ≥3 for this measure. Higher scores indicate greater perceived acceptability.
Percentage of participants who engage in at least one cycle of intervention | 6 months after the final DRV during study exit interviews [participant specific
  The percentages of participating patients, parents, and multidisciplinary clinicians who engage in at least one cycle of the intervention.

SECONDARY OUTCOMES:
Potential impact of the RIGHTimeCPV intervention on communication quality, concordance in prognostic understanding, and therapeutic alliance between patients/families and multidisciplinary clinicians | Between Day 1-30 after the CPV timepoint [participant specific], between Day 1-30 after the DRV timepoint [participant specific], and 6 months after the final DRV during study exit interviews [participant specific
  This outcome will be assessed through generation of qualitative thematic findings. Specifically, qualitative data gathered from audio-recorded encounters at the Communication Preferences Visit (CPV) and DRV timepoints, as well as post-intervention interviews, will undergo rapid qualitative analysis and reflexive thematic analysis to explore participating patient, caregiver, and clinician impressions of the intervention's impact on communication quality, prognostic understanding, and therapeutic alliance between patients/caregivers and multidisciplinary clinicians.
Whether the practice of eliciting, sharing, and honoring individualized communication preferences is sustained by clinicians after participation in the RIGHTimeCPV intervention | 6 months after the final DRV during study exit interviews [participant specific
  Through analysis of the final post-intervention interview, the investigators will generate thematic findings related to participant perspectives on the intervention's impact on individual attitudes and behaviors and whether the practice of eliciting, sharing, and honoring individualized communication preferences was sustained by clinicians after participation in the RIGHTimeCPV intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Erica C. Kaye, MD, MPH, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols